CLINICAL TRIAL: NCT03684837
Title: D Vitamine Supplementation and Whole Body Vibration Altering Functional Outcomes
Brief Title: D Vitamine and Whole Body Vibration in Functional Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maíra F Pessoa (Other)
Responsible Party: Sponsor-Investigator, Maíra F Pessoa, Clinical Professor, Universidade Federal de Pernambuco
Organization: Universidade Federal de Pernambuco (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COPDinfl
Record Dates: First submitted 2018-09-19; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: COPD; Aging
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D vitamine (Active Comparator): a dose for week
  Interventions: Dietary Supplement: Vitamine D supplementation; Other: chronic exercise in whole body vibration (WBV)
- D vitamine placebo (Placebo Comparator): a dose for week
  Interventions: Other: chronic exercise in whole body vibration (WBV)

INTERVENTIONS:
Dietary Supplement: Vitamine D supplementation — a vitamine D dose for week
  Arms: D vitamine
Other: chronic exercise in whole body vibration (WBV) — exercise in WBV during 03 months, e times per week

SUMMARY:
Older with Chronic obstructive Pulmonary Disease (COPD) were submitted to chronic whole body vibration training during 03 months, receiving a vitamine D dose for each week or placebo vitamine. This group was compared with healthy older which were submitted to the same intervention.

ELIGIBILITY:
Inclusion Criteria:

* Older patients with COPD
* Both genders
* Sedentary according to International Physical Activity Questionnaire (IPAQ) short form
* BMI in between 22.9 and 28 kg/m2.
* Older patients with COPD should have a clinical-functional diagnosis of the disease according to GOLD (GOLD, 2018), have been ex-smokers and have not used corticosteroids or have used this drug in a stable way for at least one year (without dosage or medication modifications).
* Older volunteers should be self-referenced healthy or, if they had systemic arterial hypertension or diabetes mellitus, these comorbidities should be controlled by diet or regular medication use.

Exclusion Criteria:

* Older patients with COPD who had episodes of exacerbation in the last three months, those with pulmonary rehabilitation programs in the last year, those who used home oxygen therapy, and patients with COPD-associated comorbidities were excluded.
* Volunteers of both groups who were taking vitamin D were excluded, as well as the current smokers, although occasional, volunteers with a history of labyrinthitis or thromboembolism, who had undergone surgical procedures of any size in the last year, such as plaques, pins or cardiac pacemakers, those with unconsolidated fractures that used medications that affected bone metabolism or lean mass, or those who had difficulties adapting to the assessment or the training protocol.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Functional capacity | before and immediately up to 12 weeks in WBV training.
  Change in walk distance achieved in metres, measured during the six minute walk test

SECONDARY OUTCOMES:
Balance static and dynamic | before and immediately up to 12 weeks in WBV training.
  Change in total scores of Tinetti index, composed by 16 items divided into 2 sections: static balance (9 items) with 16 points and gait or dynamic balance (7 items) with 12 points, summed in a total score of 28 points. Individuals scoring < 26 points have a risk for falling.
Gait speed | before and immediately up to 12 weeks in WBV training.
  Change in time in seconds registered in Timed Up and Go test
Body composition | before and immediately up to 12 weeks in WBV training.
  Change in electrical bioimpedance measuring the fat mass and lean mass in kilograms each one, in total body
Quality of life measure by WHOQOL | before and immediately up to 12 weeks in WBV training.
  Change in total value obtained from WHOQOL-old questionnaire (World Health Organization of Quality Of Life) that evaluate in older the domains: sensory abilities; autonomy; past, present and future activities; social participation; death & dying; and intimacy. The Quality of life needs to improve when it is 1 to 2,9; is regular 3 to 3.9 points; good between 4 up to 4.9 and very good with 5 points.
Peripheral strength | before and immediately up to 12 weeks in WBV training.
  Change in mean value obtained from 03 maneuvers of isokinetic contraction in a hand dynamometer (device that measure strength in handgrip), measured in centimeters of water.
Respiratory strength | before and immediately up to 12 weeks in WBV training.
  Change in major value obtained after 03 maneuvers in manovacuometer (device that measure manometry for expiratory pressure and vacuum generated for the inspiratory pressure), all in centimeters of water.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No